CLINICAL TRIAL: NCT01423552
Title: Correlation of Immunosuppressant Pharmacokinetics, Pharmacodynamics, Pharmacogenomics and Outcomes Following Heart Transplantation
Brief Title: Pharmacology of Immunosuppressants Following Heart Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nigel E. Drury (Other)
Responsible Party: Sponsor-Investigator, Nigel E. Drury, Specialist Registrar & Honorary Clinical Lecturer, University Hospital Birmingham
Organization: University Hospital Birmingham (Other)
Other Study IDs: RRK4220
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Heart Transplantation
Keywords: Heart transplantation; Immunosuppression; Pharmacokinetics; Pharmacogenetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Myocardial biopsy, whole blood, peripheral lymphocytes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post-heart transplant: All patients undergoing heart transplantation at the Queen Elizabeth Hosptial Birmingham in the last 12 months or in the next year.

SUMMARY:
The ongoing success of transplantation is largely due to the development of drugs to stop the patient's body from rejecting the new organ. In addition to steroids, two main types of drug are used to suppress the immune system following heart transplantation: calcineurin inhibitors (Ciclosporin-A or Tacrolimus) and mycophenolate. However, different patients respond in different ways to these drugs, with the same dose leading to different levels of the drug in the blood. This varies due to genetic and other factors such as age, kidney function and the use of other drugs. Therefore, the levels of immunosuppressive drugs in the blood are routinely measured and the dose adjusted accordingly. However, some patients still experience episodes of rejection despite apparently acceptable levels. In this study, the investigators will measure levels of the drugs (in the blood, in a type of white blood cell called T-cells and in the heart muscle) and the effectiveness of the drugs on T-cells. The investigators will compare these levels with patient genetic factors and the amount of rejection measured on heart biopsies. This will enable us to better understand how the blood and tissue levels of these drugs change with genetic and other factors in order to optimise immunosuppressive therapy and further improve outcomes from heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing heart transplantation

Exclusion Criteria:

* Decline participation
* Previous transplantation of another organ and already receiving chronic immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart transplantation at the Queen Elizabeth Hosptial Birmingham.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-11

PRIMARY OUTCOMES:
Correlation of immunosuppressant drug levels in different compartments with evidence of rejection | Multiple timepoints in first 12 months after transplantation
  We will compare the levels of the drugs in different compartments of the body (in the blood, within white blood cells and within the heart muscle itself) with how well the drugs are working ie. how well the heart is functioning and the level of rejection seen on routine heart biopsies. Drug levels will be measured at C0 (trough) and C2 (peak).

SECONDARY OUTCOMES:
Correlation of individual patient genetic and other factors with levels of immunosuppressant drugs in different compartments | Multiple timepoints in first 12 months after transplantation
  We will also compare these results with patient genetic and other factors (eg. age, kidney function, use of other drugs) to better understand how these factors affect the levels of the drugs in different compartments of the body. Drug levels will be measured at C0 (trough) and C2 (peak).

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Bonser, MD FRCS, Principal Investigator — University Hospital Birmingham
Locations (2):
- Basil Hetzel Institute for Medical Research, Adelaide, South Australia, Australia
- Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands, United Kingdom